CLINICAL TRIAL: NCT02398487
Title: Head-To-Head Comparision of Personal Vaporizers Versus Cigalike: Prospective 6-Month Randomized Control Design Study
Brief Title: Personal Vaporizer vs Cigalike
Acronym: VAPECIG 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita degli Studi di Catania (Other)
Responsible Party: Principal Investigator, Riccardo Polosa, Professor, Universita degli Studi di Catania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VAPECIG 2
Record Dates: First submitted 2014-06-09; First posted 2015-03-25 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Cigarette Addiction
MeSH Terms: interventions — Tobacco Use Cessation Devices; Nebulizers and Vaporizers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Personal Vaporizer (Active Comparator): Personal Vaporizer loaded with nicotine
  Interventions: Device: Personal Vaporizer with nicotine
- Cigalike (Active Comparator): Cigalike loaded with nicotine
  Interventions: Device: cigalike with nicotine
- Usual smoking (No Intervention)

INTERVENTIONS:
Device: cigalike with nicotine — cigalike 24 mg nicotine or 16 mg nicotine
  Arms: Cigalike
Device: Personal Vaporizer with nicotine — Personal Vaporizer 16 mg nicotine or 9 mg nicotine
  Arms: Personal Vaporizer

SUMMARY:
This is a pilot study to compare efficiency and tolerability of a personal vaporizers (PV) new generation electronic cigarette loaded with nicotine e-liquid with cigalike new generation electronic cigarette loaded with nicotine and usual smoking habits, in a group of well characterized regular smokers unwilling to quit.

DETAILED DESCRIPTION:
RATIONALE

The results of ECLAT - the first randomized controlled trial addressing the impact of electronic cigarette use in relation to smoking reduction, smoking abstinence and safety long-term - have revealed important and persistent modifications in the smoking habits of 300 smokers (not intending to quit) with significant reduction in tobacco cigarettes' consumption (1).

Surprisingly, the reduction in cig/day use in ECLAT was not much different among study groups, with the non-nicotine study group performing much like both high and low nicotine study groups. This was because, with the products used in ECLAT, saliva cotinine levels were well below the concentration threshold considered to be representative for regular smokers (2) or experienced electronic cigarette users (3) in both high and low nicotine study groups. Specifically, the model under investigation in ECLAT is not very efficient at delivering nicotine (4).

With this in mind, we have designed a pilot study to compare efficiency and tolerability of a personal vaporizers (PV) new generation electronic cigarette loaded with nicotine e-liquid with cigalike new generation electronic cigarette loaded with nicotine and usual smoking habits, in a group of well characterized regular smokers unwilling to quit.

STUDY OBJECTIVES

Aims of this pilot study are:

* to assess if a Personal Vaporizers (PV) can effectively reduce tobacco smoking
* to compare if efficacy data with PV E-cigs are better than "cigalike" efficacy
* to evaluate if PV E-cigs are safe to use

METHODS

Study Population 200 regular smokers (smoking ≥ 10 cigarettes per day for at least the past 5 years; eCO ≥ 10 ppm), with an age of 18-70 years, in good general health; and committed to follow the trial procedures will be recruited following placement of advertisements in local newspapers and radio/TV network. Exclusion criteria will include: recent vaping history (stopped vaping less than 3 months ago); use of any other form of non combustible nicotine containing products (chewable tobacco or nicotine replacement therapy) symptomatic cardiovascular disease; clinical history of asthma and chronic obstructive pulmonary disease (COPD); regular psychotropic medication use; current or past history of alcohol abuse; use of smokeless tobacco or nicotine replacement therapy, and pregnancy or breastfeeding.

Study Products

Personal Vaporizer electronic cigarette This new generation device consist of a large lithium battery part (capacity of 2600 mAh) with an internal electronic circuit which includes a current stabilizer and allows the user to manually adjust the energy applied to the atomizer. A new-generation atomizer will be used and will be filled with approximately 2 ml of liquid. The Energy delivery to the atomizer will be set to 9 watts.

These electronic cigarettes will be provided free of charge by the manufacturer.

The liquid will be provided free of charge by the manufacturer Alterna Farmaceutici, Francia Farmaceutici group.

"Cigarette-like Electronic Cigarette" The Cigalike e-Cigarette is a disposable battery-powered electronic nicotine delivery device (ENDD) - that closely resembles the shape of a tobacco cigarette - designed for the purpose of nicotine (and/or aroma) delivery, where no tobacco or combustion is necessary for its operation. This e-Cigarette contains a propylene glycol-free liquid consisting of distilled water, FCC grade vegetable glycerin, natural flavors, artificial flavors, citric acid and may also contain pharmaceutical grade nicotine. The lithium battery has a capacity of 250 mAh and will be fully charged before use. Cartomizers will be filled with approximately 1 ml of a nicotine containing liquid.These electronic cigarettes will be provided free of charge by the manufacturer.

Study Design and Procedures Two hundred regular smokers, (not willing to quit) will be recruited in our center following placement of advertisements in local newspapers and radio/TV network. At baseline, participants will be randomized into three separate study groups. Fifty participants randomized in study group A will receive a "Personal Vaporizer electronic cigarette" and 24-weeks supply of e-liquid (active group); fifty subjects in study group B, 24-week supply of "Cigarette-like Electronic Cigarette" (active group); one hundred participants in study group C will continue usual smoking (control group).

Study Schedule Participants will attend their study visits at the smoking cessation clinic at approximately the same time of day. With the exception of the baseline study day, most visits will take approximately 10-15 minutes.

At baseline (study visit 1), socio-demographic factors, a detailed smoking history and craving will be annotated and individual pack-years (pack/yrs) calculated. Eligible participants will be invited to sign an informed consent form. Cigarette dependence will be measured by Fagerstrom Test for Cigarette Dependence (FTCD). Additionally, levels of carbon monoxide in exhaled breath (eCO) will be measured using a portable device (Micro CO, Micro Medical Ltd, UK). Vital signs (HR and BP), body weight, and adverse events will be also recorded at baseline.

Participants in group A and B will be given a free supply of electronic smoking (on average 2-week supply of ecigs) and instructed on how to correctly use them. Key troubleshooting support will be provided and phone numbers will be supplied for medical assistance. They will also be requested to fill a 2-weeks' study diary recording adverse events. No emphasis on encouragement, motivation and reward for the smoking cessation effort will be provided since this study was intended to monitor smokers (unwilling to quit) using in three different situations.

Baseline visit (Visit 1) in brief

* Informed consent
* Inclusion/exclusion criteria
* CRF (smoking Hx, FTND, eCO, HR, BP, weight, AEs)
* Craving/VAS
* Randomization into either study group A (with Nic) or B (no Nic)
* Provide PV Ecig or Cigalike and dispense 2-weeks supply of electronic smoking (depending on the study arm allocation)
* Dispense 2-weeks' study diary for AEs

By and large, at week-2 (study visit 2), week-4 (study visit 3), week-8, week-12, and week-24, participants will a) receive further study diaries for the residual study periods, b) have their eCO levels and vital signs recorded, c) return their completed study diaries and used study products. Additionally, saliva samples will be collected at week-12 and at week-24 for cotinine measurement in those who stated they had not smoked (not even a puff) and with an eCO ≤ 7ppm. Cotton rolls will be placed into polypropylene tubes and stored at -20°C until use. Saliva samples will be analysed in duplicate for cotinine analysis by gas chromatography. At the end of week-24 study visit, no more products will be provided by the investigators.

Week-2 visit (Visit 2) in brief

* Collect 2-weeks' study diary for AEs
* CRF (no. cig/day, eCO, HR, BP)
* Craving/VAS
* Smokers' product preference survey
* Dispense next 2-weeks supply of electronic smoking (depending on the study arm allocation)
* Dispense next 2-weeks' study diary for AEs

Week-4/8 visit (Visits 3 and 4) in brief

* Collect study diary for AEs
* CRF (no. cig/day, eCO, HR, BP)
* Craving/VAS
* Dispense next 4-weeks supply of electronic smoking (depending on the study arm allocation)
* Dispense next 4-weeks' study diary for AEs

Week-12 visit (Visit 5) in brief

* Collect study diary for AEs
* CRF (no. cig/day, eCO, HR, BP and weight)
* Craving/VAS
* Collect saliva sample* (only in those with zero cig/day and eCO ≤ 7ppm, * Times of saliva sampling requires standardization, e.g. same time of the day, within 2 hrs from last vape)
* Dispense next 12-weeks supply of electronic smoking (depending on the study arm allocation)
* Dispense next 12-weeks' study diary for AEs

Week-24 visit (Visit 6)

* Collect study diary for AEs
* CRF (physical examination, no. cig/day, eCO, HR, BP and weight)
* Craving/VAS
* Collect saliva sample* (only in those with zero cig/day and eCO ≤ 7ppm, * Times of saliva sampling requires standardization, e.g. same time of the day, within 2 hrs from last vape)
* Smokers' product preference survey

Study Outcome Measures A ≥50% reduction in the number of cig/day from baseline, defined as self-reported reduction in the number of cig/day (≥50%) compared to baseline (together with an eCO levels reduction, to objectively document a reduction from baseline), will be calculated at each study visit ("reducers").

Abstinence from smoking, defined as complete self-reported abstinence from tobacco smoking - not even a puff (together with an eCO concentration of ≤7 ppm), will be calculated at each study visit ("quitters"). Failing to meet the above criteria defines smoking reduction/cessation failure.

Adverse events, symptoms thought to be related to tobacco smoking and e-Cigarette use and to withdrawal from nicotine will be annotated at baseline and at each subsequent study visit on the adverse event page of the study diary. Vital signs will be also recorded. Participants' perception and liking of the product will be assessed by asking to rate their level of satisfaction with the products compared to their own cigarettes using a visual analogue scale (VAS) from 0 to 10 points (0 = being 'completely unsatisfied', 10 being = 'fully satisfied'); using the same scale, they will also rate how much they miss their own brand (0 = being 'did not miss it at all', 10 being = 'missed too much') and whether they would recommend it to a friend/relative (0 = being 'not recommended at all', 10 being = 'absolutely recommended').

ELIGIBILITY:
Inclusion Criteria:

* in good general health
* committed to follow the trial procedures

Exclusion Criteria

* recent vaping history (stopped vaping less than 3 months ago)
* use of any other form of non combustible nicotine containing products (chewable tobacco or nicotine replacement therapy) symptomatic cardiovascular disease
* clinical history of asthma and chronic obstructive pulmonary disease (COPD)
* regular psychotropic medication use
* current or past history of alcohol abuse
* use of smokeless tobacco or nicotine replacement therapy, and pregnancy or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Smoking Reduction | 24 week
  50% reduction of cigarette smoked compared to baseline

SECONDARY OUTCOMES:
Smoking Cessation | 24 week
  complete abstinence

CONTACTS AND LOCATIONS:
Locations (1):
- Centro per la Prevenzione e Cura del Tabagismo University of Catania, Catania, Catania, Italy